CLINICAL TRIAL: NCT01900522
Title: A Phase 1, Randomized, Placebo- Controlled, Double-Blind Safety, Tolerability, Pharmacokinetic, and Exploratory Pharmacodynamic Study in Healthy Subjects and Subjects With Stable Schizophrenia After Multiple Doses of ITI-214
Brief Title: Safety and Tolerability of Multiple Doses of ITI-214 in Healthy Adults and in Adults With Stable Schizophrenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision; No Safety or Efficacy Concerns
Sponsor: Takeda (Industry)
Collaborators: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: ITI-214_102; U1111-1142-0234 (Registry Identifier: UTN (WHO))
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia
Keywords: Drug therapy
MeSH Terms: conditions — Schizophrenia | interventions — Aging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multiple Rising Dose (MRD) Phase: Ascending ITI-214 Doses (Experimental): ITI-214 Doses (A, B, C, D, matching placebo), solution, orally, once daily for 14 days.
  Interventions: Drug: ITI-214 Dose A; Drug: ITI-214 Dose B; Drug: ITI-214 Dose C; Drug: ITI-214 Dose D (Elderly); Drug: Placebo
- Neuroimaging Phase: ITI-214 Doses (Experimental): ITI-214 (E,F, G, H, matching Placebo) Oral solution, once daily for 7 days in 3 periods with placebo and two of the ITI-214 Doses (E, F, G and H) in a cross-over fashion with minimum 7 days washout between periods
  Interventions: Drug: ITI-214 Dose E; Drug: ITI-214 Dose F; Drug: ITI-214 Dose G; Drug: ITI-214 Dose H; Drug: Placebo

INTERVENTIONS:
Drug: ITI-214 Dose A — ITI-214 Dose A Oral Solution
  Arms: Multiple Rising Dose (MRD) Phase: Ascending ITI-214 Doses
Drug: ITI-214 Dose B — ITI-214 Oral Solution Dose B
  Arms: Multiple Rising Dose (MRD) Phase: Ascending ITI-214 Doses
Drug: ITI-214 Dose C — ITI-214 Dose C Oral Solution
  Arms: Multiple Rising Dose (MRD) Phase: Ascending ITI-214 Doses
Drug: ITI-214 Dose D (Elderly) — ITI-214 Dose D (Elderly) Oral Solution
  Arms: Multiple Rising Dose (MRD) Phase: Ascending ITI-214 Doses
Drug: Placebo — ITI-214 Matching Placebo Oral Solution
  Arms: Multiple Rising Dose (MRD) Phase: Ascending ITI-214 Doses
Drug: ITI-214 Dose E — ITI-214 Dose E Oral Solution
  Arms: Neuroimaging Phase: ITI-214 Doses
Drug: ITI-214 Dose F — ITI-214 Dose F Oral Solution
  Arms: Neuroimaging Phase: ITI-214 Doses
Drug: ITI-214 Dose G — ITI-214 Dose G Oral Solution
  Arms: Neuroimaging Phase: ITI-214 Doses
Drug: ITI-214 Dose H — ITI-214 Dose H Oral Solution
  Arms: Neuroimaging Phase: ITI-214 Doses
Drug: Placebo — ITI-214 Matching Placebo Oral Solution
  Arms: Neuroimaging Phase: ITI-214 Doses

SUMMARY:
The purpose of this study is to characterize the safety and tolerability profile of ITI-214 when administered as multiple doses of oral solution at escalating dose levels.

DETAILED DESCRIPTION:
The drug being tested in this study is called ITI-214. This study will look at how well different doses of ITI-214 are tolerated in healthy people and in people with stable schizophrenia. In addition, exploratory neuroimaging will be conducted in participants with schizophrenia.

This multi-center trial will be conducted in the United States. The study will be comprised of 2 parts: Multiple-Rising Dose (MRD) and Neuroimaging (NI). Approximately 40 healthy participants are planned to be enrolled in the MRD part of the study and approximately 36 patients with stable schizophrenia are planned to be enrolled in the Neuroimaging part of the study.

Participants in the MRD (parallel design) part will be enrolled in cohorts for different dose levels. In each dose cohort, participants will be randomly assigned to active dose or placebo-which will remain undisclosed to participants and study doctor during the study (unless there is an urgent medical need). The following dose cohorts will be enrolled: Doses A, B, C, and D.

Participants will be asked to take the study drug in oral solution once daily for a total of 14 days while confined at the study site. Participants will be contacted by telephone 22 and 44 days after last dose of study drug for a follow-up assessment.

Participants in the Neuroimaging (NI) part of the study will be randomly assigned to one of six treatment sequences. Each sequence consists of 3 cross-over treatment periods. The following doses will be tested: Doses E, F, G, and H.

Each participant will undergo 3 treatment periods of placebo or ITI-214 once daily dosing for 7 days in each of the periods. There will be a washout period of a minimum of 7 days between treatment periods. Participants will be confined at the study site for 5 days of each treatment period and will report to the site on other dosing days for study drug administration. There will be follow-up assessments on Days 14 and 37 of Period 3.

Study was terminated due to business decision. The study compound is being transferred to Intra-Cellular Therapies, Inc.

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants

1. Is capable of understanding and complying with protocol requirements.
2. The participant or; when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is a healthy man or woman, aged 18 to 55 years, inclusive (non-elderly) or aged ≥65 years (elderly), at the time of informed consent and first study medication dose.
4. Weighs at least 50 kg and has a body mass index (BMI) between 18.0 and 35.0 kg/m^2, inclusive at Screening.
5. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
6. A female participant with no childbearing potential. The participant has been surgically sterilized (hysterectomy, bilateral oophorectomy or tubal ligation) or who are postmenopausal (defined as continuous amenorrhea of at least 2 years and follicle-stimulating hormone (FSH) >40 IU/L.

Participants with schizophrenia:

1. Is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is capable of consenting. A standard evaluation by a psychiatrist will be implemented to assess the participant's capacity to consent.
4. Is a man or woman, aged 18 to 60 years (non-elderly), inclusive, or aged ≥65 years (elderly, if decided to enroll), at the time of informed consent and first study medication dose.
5. Weighs at least 50 kg and has a body mass index (BMI) between 18.0 and 35.0 kg/m^2, inclusive at Screening.
6. Is diagnosed with schizophrenia criteria as defined by the Diagnostic & Statistical Manual of Mental Disorders 4th Edition - Text Revision (DSM-IV-TR) and determined by the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I), schizoaffective disorder, or schizophreniform disorder; on a stable dose of one and only one of the second generation antipsychotics (except olanzapine, clozapine, or quetiapine) for at least 2 months by medical history and assessed by site staff; Positive and Negative Syndrome Scale (PANSS) Conceptual Disorganization item score ≤ 4 and PANSS Hallucinatory Behavior or Unusual Thought Content item scores ≤ 4. For the MRD part, the subject is diagnosed with schizophrenia criteria as defined by the DSM-IV-TR and determined by the SCID-I, schizoaffective disorder, or schizophreniform disorder; on a stable dose of one and only one of the second generation antipsychotics (except clozapine) for at least 2 months by medical history and assessed by site staff; PANSS Conceptual Disorganization item score ≤ 4 and PANSS Hallucinatory Behavior or Unusual Thought Content item scores ≤ 4.
7. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
8. A female subject of childbearing potential* who is sexually active with a nonsterilized* male partner agrees to use an acceptable method of contraception* from signing of informed consent and for 12 weeks postdose.

Exclusion Criteria:

Healthy Participants

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Has received ITI-214 in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a known hypersensitivity to any component of the formulation of ITI-214 or Listerine.
6. Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -1).
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
8. Has taken any excluded medication, supplements, or food products.
9. Is pregnant or lactating or intending to become pregnant before, during, or within 12 weeks after participating in this study; or intending to donate ova during such time period.
10. If male, the participant intends to donate sperm during the course of this study or for 12 weeks after last dose.
11. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking ITI-214, or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias. Elderly participants may have been eligible for enrollment if approved by the investigator and Takeda medical monitor.
12. Has mental retardation or medical condition that can cause cognitive impairment.
13. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, any surgical intervention known to impact absorption [eg, bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent [more than once per week] occurrence of heartburn).
14. Has a history of cancer, except basal cell carcinoma which has not been in remission for at least 5 years prior to Check-in (Day -1)
15. Has a positive test result for hepatitis B surface antigen (HBsAg), antibody to hepatitis C (anti-HCV) or a known history of human immunodeficiency virus infection at Screening.
16. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -1). Cotinine test is positive at Screening or Check-in (Day -1). The participant has poor peripheral venous access.
17. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days prior the first dose of study medication.
18. Has a Screening or Check-in (Day -1) abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved and documented by signature by the principal investigator.
19. Has a supine blood pressure outside the ranges of 90 to 140 mm Hg for systolic and 60 to 90 mm Hg for diastolic, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1).
20. Has a resting heart rate outside the range 50 to 100 bpm, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1).
21. Has a QTcF >440 ms (males) or >460 ms (females) or PR outside the range 120 to 220 ms, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1).
22. Has abnormal Screening or Check-in (Day -1) laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 the upper limits of normal.
23. Has a risk of suicide according to the Investigator's clinical judgment (eg, per Columbia-Suicide Severity Rating Scale [C-SSRS] or has made a suicide attempt in the previous 6 months).

Participants with schizophrenia:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
3. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine disease, or psychiatric disorder, or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
4. Has a known hypersensitivity to any component of the formulation of ITI-214 or Listerine.
5. Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -2 of Periods 1).
6. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
7. Has taken any excluded medication, supplements, or food products.
8. Iis pregnant or lactating or intending to become pregnant before, during, or within 12 weeks after participating in this study; or intending to donate ova during such time period.
9. If male, the participant intends to donate sperm during the course of this study or for 12 weeks after last dose.
10. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking ITI-214, or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
11. Has mental retardation.
12. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, any surgical intervention known to impact absorption [eg, bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent [more than once per week] occurrence of heartburn).
13. Subject has a history of cancer, except basal cell carcinoma which has not been in remission for at least 5 years prior to Check-in Day -1 for MRD part) and Day -2 of Period 1 for Neuroimaging part ).
14. Has a positive test result for hepatitis B surface antigen (HBsAg), antibody to hepatitis C (anti-HCV) or a known history of human immunodeficiency virus infection at Screening.
15. Participants who currently use nicotine-containing products but will not maintain their nicotine use habit throughout the study.
16. Has poor peripheral venous access.
17. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days prior the first dose of study medication.
18. The subject has a Screening or Check-in (Day -1 for MRD part) and Check-in (Day -2 of Period 1 for Neuroimaging part) abnormal (clinically significant) ECG. Entry of any subject with an abnormal (not clinically significant) ECG must be approved and documented by signature by the principal investigator or medically qualified sub-investigator.
19. The subject has a supine blood pressure outside the ranges of 90 to 140 mm Hg for systolic and 60 to 90 mm Hg for diastolic, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1 for MRD part) and Check-in (Day -2 of Period 1 for Neuroimaging part).
20. The subject has a resting heart rate outside the range 50 to 100 bpm, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1 for MRD part) and Check-in (Day -2 of Period 1 for Neuroimaging part).
21. The subject has a QTcF >440 ms (males) or >460 ms (females) or PR outside the range 120 to 220 ms, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1 for MRD part) and Check-in (Day -2 of Period 1 for Neuroimaging part).
22. The subject has abnormal Screening or Check-in (Day -1 for MRD part) and Check-in (Day -2 of Period 1 for Neuroimaging part) laboratory values that suggest a clinically significant underlying disease or has the following lab abnormalities: ALT and/or AST >1.5 the upper limits of normal.
23. Has a risk of suicide according to the Investigator's clinical judgment (eg, per C-SSRS) or has made a suicide attempt in the previous 6 months.
24. Has a current diagnosis of significant psychiatric illness other than schizophrenia, per DSM-IV.
25. For subjects enrolled in the neuroimaging part at the site performing fMRI, the subject has a personal history of claustrophobia or inability to tolerate mock scanner environment during habituation/screening session; surgery involving metal implants, non-removable body metal objects (metal body piercing, dentures, dental plates or bridges, any implanted device that is electrically, magnetically, and mechanically activated); a personal history of seizures, other neurologic disease, or increased intracranial pressure; history of open head injury or significant closed head injury; or hearing loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who experience at least one treatment-emergent adverse event (TEAE) | Day 1 to Day 44 (up to 24 hours postdose)
  A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug and within 30 days after receiving the last dose of study drug. A TEAE may also be a pre-treatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug, which increases in intensity after the start of dosing.

SECONDARY OUTCOMES:
Tmax: Time to Reach the Maximum Plasma Concentration | Days 1 and 14 (up to 24 hours postdose)
  Time to reach the maximum observed plasma concentration for ITI-214F and ITI-214F metabolite IC200338 after a single dose (Day 1) and multiple dosing (Day 14).
Cmax: Maximum Observed Plasma Concentration | Days 1 and 14 (up to 24 hours postdose)
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Cmax will be measured for ITI-214F and ITI-214F metabolite IC200338 after a single dose (Day 1) and multiple dosing (Day 14).
AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration | Days 1 and 14 (up to 24 hours postdose)
  AUC(0-tlqc) is a measure of total plasma exposure to a drug from time 0 to time of the Last Quantifiable Concentration and will be measured for ITI-214F and ITI-214F metabolite IC200338 after a single dose (Day 1) and multiple dosing (Day 14).
AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose | Days 1 and 14 (up to 24 hours postdose)
  AUC(0-24) is a measure of total plasma exposure to the drug from Time 0 to 24 hours post-dose for ITI-214F and ITI-214F metabolite IC200338 after a single dose (Day 1) and multiple dosing (Day 14).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Glendale, California
  - New York, New York